CLINICAL TRIAL: NCT01286532
Title: A Six-month Non-interventional Prospective Study of Various Controller Therapies for Moderate Persistent and Severe Persistent Asthma in Children in Real Life Outpatient Clinical Practice
Brief Title: Asthma in Children
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RRU-XXX-2010/1
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
Keywords: Asthma, Asthma in Children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children (male or female) aged 5 to 11 years inclusive on step 3 asthma combination therapy with ICS(inhalation glucocorticosteroids) and LABA ( long-acting b2-agonist) who have completed at least one valid CACT assessment after the study entry

SUMMARY:
This is a six-month non-interventional prospective study of various controller therapies in children with asthma in outpatient clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Child (male or female) aged 5 to 11 years inclusive
* Provision of Subject Informed Consent Form for anonymous data collection and their subsequent use (must be signed by any of the parents)
* The child must be included in an out-patient observation program at a medical institution for established bronchial asthma diagnosis for at least 1 year prior to enrolment and diagnosed with moderate to severe bronchial asthma at the time of enrolment
* The child must have at least one documented bronchial asthma exacerbation in previous 1 year (including hospital admissions for bronchial asthma exacerbations, any cases of daytime hospital treatment without overnight stays and any cases of oral administration of glucocorticoids on an out-patient basis for > 3 consecutive days)
* Out-patient receiving step 3 controller treatments with fixed dose combinations of ICSs and LABA or treatment with separate administration of glucocorticoids and LABA in stable doses with adequate control of bronchial asthma symptoms
* The patient administered with short-acting β2 agonists (inhalational) or rapidly released methylxanthines (oral) in the doses approved for the respective age as a rescue on-demand therapies during the preceding month

Exclusion Criteria:

* Cystic fibrosis, α1-antitrypsin deficiency or congenital abnormalities of lung development
* Severe comorbidities affecting the patient's overall performance
* In the physician's opinion, the patient is not able to comply with the protocol requirements
* Expected specific hyposensibilization within next 6 months
* Expected treatment at health resort facilities within next 6 months
* Other reasons that in the physician's opinion will prevent reliable assessments of the study treatment efficacy

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children (male or female) aged 5 to 11 years inclusive on step 3 asthma combination therapy with ICS and LABA who have completed at least one valid CACT assessment after the study entry
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To compare percentage (%) of responding children by the end of 6-month observation. Responders are defined as children with adequate control of symptoms at the end of 6 months observation (Childhood Asthma Control Test (CACT) score > 19) | 3 visits for 6 month

SECONDARY OUTCOMES:
To determine mean number of severe bronchial asthma exacerbations within 6 months | 3 visits for 6 month
To determine mean duration of bronchial asthma exacerbations including hospital admissions, daytime hospital treatment and any cases of oral administration of glucocorticoids > 3 consecutive days during the observation period | 3 visits for 6 month
To determine mean requirement in short-acting β2-agonists and/or rapidly released methylxanthines per week during the period of observation | 3 visits for 6 month
To determine the independent factors associated with failure of treatment of asthma (demographic and baseline patient data, site) | 3 visits for 6 month

CONTACTS AND LOCATIONS:
Locations (11):
- Russia (11):
  - Research site, Chelyabinsk
  - Research site, Moscow
  - Research site, N.Novgorod
  - Research site, Novosibirsk
  - Research site, Rostov-on-Don
  - Research site, Saint Petersburg
  - Research site, Samara
  - Research site, Tula
  - Research site, Tver'
  - Research site, Ufa
  - Research site, Volgograd